CLINICAL TRIAL: NCT05350592
Title: Low-dose Dobutamine Infusion and Single-dose Tocilizumab in Acute Myocardial Infarction Patients With High Risk of Cardiogenic Shock Development - a 2x2 Multifactorial, Double-blinded, Randomized, Placebo Controlled Trial
Brief Title: Low-Dose Dobutamine and Single-Dose Tocilizumab in Acute Myocardial Infarction With High Risk of Cardiogenic Shock
Acronym: DOBERMANN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry); Simon Spies Fonden (Unknown); Helge Peetz og Verner Peetz og hustru Vilma Peetz Legat (Unknown)
Responsible Party: Principal Investigator, Helle Søholm, MD, PhD, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-CARD-Pharma001; 2021-002028-19 (EudraCT Number); H-21045751 (Registry Identifier: National Committee on Health Research Ethics); U1111-1277-8523 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2022-03-08; First posted 2022-04-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Acute Myocardial Infarction; Cardiogenic Shock
Keywords: acute myocardial infarction; cardiogenic shock; AMI; inflammation; proBNP; AMI-CS; infarct size; STEMI
MeSH Terms: conditions — Shock, Cardiogenic; Inflammation; ST Elevation Myocardial Infarction | interventions — tocilizumab; Dobutamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 2x2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tocilizumab + Dobutamine (Active Comparator): Tocilizumab IV 280 mg (100mL/hour, 1 hour) Dobutamine IV 5 micrograms/kg/minute (5mL/hour, 24 hours)
  Interventions: Drug: Tocilizumab; Drug: Dobutamine
- Tocilizumab + Placebo (Active Comparator): Tocilizumab IV 280 mg (100mL/hour, 1 hour) NaCl 0,9% IV (5mL/hour, 24 hours)
  Interventions: Drug: Tocilizumab; Drug: NaCl 0.9%
- Placebo + Dobutamine (Active Comparator): NaCl 0,9% IV (100mL/hour, 1 hour) Dobutamine IV 5 micrograms/kg/minute (5mL/hour, 24 hours)
  Interventions: Drug: Dobutamine; Drug: NaCl 0.9%
- Placebo + Placebo (Placebo Comparator): NaCl 0,9% IV (100mL/hour, 1 hour) NaCl 0,9% IV (5mL/hour, 24 hours)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Tocilizumab — Single bolus
  Other Names: RoActemra (Actemra)
  Arms: Tocilizumab + Dobutamine; Tocilizumab + Placebo
Drug: Dobutamine — Continous weight-adjusted infusion
  Other Names: Dobutrex
  Arms: Placebo + Dobutamine; Tocilizumab + Dobutamine
Drug: NaCl 0.9% — Placebo comparator and diluent
  Other Names: Saline isotonic
  Arms: Placebo + Dobutamine; Placebo + Placebo; Tocilizumab + Placebo

SUMMARY:
In the present study, we aim to investigate the effects of dobutamine infusion and/or a single intravenous (IV) dose of the IL-6 antagonist Tocilizumab administered after percutaneous coronary intervention (PCI) to patients with acute myocardial infarction (AMI) presenting < 24 hours from onset of chest pain and an intermediate to high risk of cardiogenic shock (CS) by assessment with the ORBI risk score (≥10 - not in overt shock at hospital admission).

Plasma concentrations of pro-B-type natriuretic peptide (proBNP) as a proxy for development of cardiogenic shock (CS) and hemodynamic instability will be sampled for primary endpoint analysis.

Effects on clinical parameters, mortality, morbidity as well as specific indicators of inflammation, cardiac function, and infarct size will secondarily be assessed noninvasively.

The rationale behind the current study is that inflammatory and neurohormonal responses are associated with subclinical hemodynamic instability in patients with AMI with high risk of CS have worse outcomes. The potentially unstable condition may be targeted pharmacologically as an add-on to existing therapy. This is investigated in patients at elevated risk of CS by sampling biomarkers reflecting the inflammatory and neurohormonal responses, as well as determining effects on patient outcomes and infarct size.

DETAILED DESCRIPTION:
The planned study is an investigator-initiated, randomized, double blinded clinical trial.

Consecutive patients at Copenhagen University Hospital, Rigshospitalet admitted with AMI < 24 hours from chest pain will be screened.

Patients eligible for trial inclusion will be randomized 2:2 to receive a continuous IV dobutamine infusion of 5 mcg/kg/minute versus placebo for 24 hours and to receive a single IV dose of tocilizumab (1-hour infusion) versus placebo administered after PCI.

Treatment with the investigational drug will be initiated as soon as possible but no later than 2 hours after transfer to the coronary care unit (CCU) and after informed consent. All included patients will follow usual treatment according to current guidelines.

The biomarker proBNP will be measured in blood samples drawn upon hospital admission in patients with ORBI risk score ≥10, and after 12, 24, 36 and 48 hours from admission.

After treatment termination, 2D-echocardiography will be performed acutely and within 2 days to evaluate left ventricular ejection fraction (LVEF), and cardiac magnetic resonance imaging (cMRi) with late gadolinium enhancement technique prior to hospital discharge as close to 48 hours post-MI and after 3 months after discharge will be performed to calculate area at risk and salvage index after AMI.Blood samples (40 mL) will be obtained and stored in a biobank for subsequent measurement of biomarkers reflecting inflammation, neurohormonal activation, neuronal injury, connective tissue function and other relevant pathophysiological processes.

These biomarkers will solely have research interest and no clinical implications. Furthermore, no genetic biomarkers and markers associated with malignancy development will be measured. Any leftover blood from the research biobank will be transferred to a biobank for future research and stored for up to 10 years solely for research purposes. After this period blood samples will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Revascularization with PCI
* Presentation within 24 hours of chest pain
* ORBI risk score ≥ 10
* Age ≥ 18

Exclusion Criteria:

* Unwilling to give informed consent to study participation
* Unable to give consent due to language barrier
* Comatose after cardiac arrest
* Cardiogenic shock with systolic blood pressure < 100 mmHg for more than 30 minutes or need for vasopressor to maintain blood pressure and arterial lactate > 2,5 (2,0) mmol/L developed before leaving the cath. lab.
* Other major clinical non-coronary condition (stroke, sepsis etc.), which can explain a high ORBI risk score
* Referral for acute coronary artery bypass grafting (CABG) (< 24 hours) after the CAG
* Contraindications against dobutamine infusion (sustained ventricular tachycardia prior to admission or noted in the cath.lab., known pheochromocytoma, idiopathic hypertrophic subaortic stenosis)
* Tocilizumab allergy
* Pregnant- or breastfeeding women
* Known liver disease/dysfunction
* Ongoing uncontrollable infection
* Immune deficiency/treatment with immunosuppressants
* Known, uncontrolled gastrointestinal (GI) disease predisposing to GI perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
ProBNP | 48 hours
  ProBNP plasma concentration being assessed at multiple time points (including the primary endpoint) will be analyzed by application of a linear mixed model of covariance. As the biomarker will be measured prior to initiation of the study drug, the models will be baseline corrected (i.e., constrained linear mixed models, CLMM). The main result of these analyses will be the treatment-by-time interaction as a marker of whether the proBNP levels change differently over time in the treatment versus the placebo arm.

SECONDARY OUTCOMES:
CS and/or cardiac arrest | Index admission
  Number of patients developing in-hospital CS and/or in-hospital cardiac arrest
Acute Infarct Size | Admission
  Magnetic-resonance imaging-estimated infarct size
Post-infarction Salvaged Myocardium | 3 months
  Magnetic-resonance imaging-estimated infarct size
Additional biomarkers | Index admission
  Reflecting neurohormonal activation, endothelial function/damage, inflammation (pro- and anti-inflammatory processes - including IL-6 and C-reactive peptide (CRP)), connective tissue damage, organ dysfunction, and other relevant physiological processes
Post-procedure assessment | Index admission
  Survey of PCI operator's post-procedure clinical assessment of the patient's survival at discharge (yes/no)
Development of non-cardiac arrest arrythmia | Index admission
  Number of patients and number of per-patient episodes of sustained ventricular tachycardia or atrial fibrillation with a frequency above 120 for more than 30 minutes
2D echocardiographic measurements of hemodynamics | Admisson, 3 months
  VTI and left ventricular function including strain measurements according to protocol
Re-admission | One year
  Number of all cause and cardiovascular admissions during the first year after index hospitalization
Heart Quality of Life (HeartQoL) | Admission, 3 months
  Heart-specific Quality of Life Questionnaire
EuroQol Group EQ-5D Quality of Life (EQ-5D-5L) | Admission, 3 months
  Quality of Life Questionnaire
HADS (Hospital Anxiety and Depression Scale) | Admission, 3 months
  In-patient Anxiety and Depression Questionnaire
The Montreal Cognitive Assessment (MOCA) | Admission, 3 months
  Clinician-administered Cognitive Test
Clinical Frailty Scale (CFS) | Admission, 3 months
  Clinician-administered Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Helle Søholm, MD, PhD, Principal Investigator — Dept. of Cardiology, Rigshospitalet; Martin Frydland, MD, PhD, Principal Investigator — Dept. of Cardiology, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data is planned to be available upon reasonable request via the Principal Investigator pending final, complete publication of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Access and final IPD criteria is pending final, complete publication of the study.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Holle SLD, Kunkel JB, Hassager C, Pecini R, Wiberg S, Palm P, Holmvang L, Bang LE, Kjaergaard J, Thomsen JH, Engstrom T, Moller JE, Lonborg JT, Soholm H, Frydland M. Low-dose dobutamine in acute myocardial infarction with intermediate to high risk of cardiogenic shock development (the DOBERMANN-D trial): study protocol for a double-blinded, placebo-controlled, single-center, randomized clinical trial. Trials. 2024 Oct 30;25(1):731. doi: 10.1186/s13063-024-08567-y. PMID 39478521
- [Background] Kunkel JB, Holle SLD, Hassager C, Pecini R, Wiberg S, Palm P, Holmvang L, Bang LE, Kjaergaard J, Thomsen JH, Engstrom T, Moller JE, Lonborg JT, Frydland M, Soholm H. Interleukin-6 receptor antibodies (tocilizumab) in acute myocardial infarction with intermediate to high risk of cardiogenic shock development (DOBERMANN-T): study protocol for a double-blinded, placebo-controlled, single-center, randomized clinical trial. Trials. 2024 Nov 5;25(1):739. doi: 10.1186/s13063-024-08573-0. PMID 39501388

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05350592/Prot_SAP_001.pdf